CLINICAL TRIAL: NCT02959632
Title: Animal Assisted Therapy Intervention for Hospitalized Patients in a Tertiary Care Center: A Pilot Study
Brief Title: Animal Assisted Therapy Intervention for Hospitalized Patients in a Tertiary Care Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ying Ying (Christina) Chen, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-007730
Record Dates: First submitted 2016-11-04; First posted 2016-11-09 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Hospitalized Patients
MeSH Terms: interventions — Animal Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients receiving AAT (Experimental): Hospitalized patients receiving Animal Assisted Therapy (AAT).
  Animal Assisted Therapy (Pet Visit) will be provided to the hospitalized patients.
  Interventions: Behavioral: Animal Assisted Therapy

INTERVENTIONS:
Behavioral: Animal Assisted Therapy — Animal Assisted Therapy is the program where a pet, usually dog will visit and interact with the patients.

SUMMARY:
The purpose of this study is to evaluate the common symptoms leading to an Animal Assisted Therapy consult, and to measure its (AAT) influence on the symptoms and feelings of hospitalized patients.

DETAILED DESCRIPTION:
Animal Assisted Therapy is being provided by the Caring Canines program and is formally available to patients by referrals. In this study, we would like to capture why patients are being referred and to measure the influence of AAT on the symptoms and feelings of patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (Patients):

* Patients admitted to St Mary's or Methodist Hospital and subsequently referred for AAT.
* Subjects undergoing Animal Assisted Therapy as part of their standard care.
* Patients 18-80 years of age.
* Patients who are able to read and answer pre and post intervention survey questionnaire and satisfaction survey.

Inclusion Criteria (Care Team Members):

* Care team members of the study participants.
* 18-80 years of age.
* Who are able to read and answer pre and post intervention survey questionnaire and satisfaction survey.

Exclusion Criteria:

Exclusion Criteria (Patients):

* Patients with diagnoses of bipolar disorder, schizophrenia or dementia.
* Unable to give consent.
* Pregnant women (as verbalized by participant).

Exclusion Criteria (Care Team Members):

* Care team members of the study participants who do not want to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11; Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Number of patients scoring improvement of symptoms using the VAS (visual analogue scale) | Baseline to 45 minutes
  We will record the number of patients scoring improvement of symptoms using the VAS (visual analogue scale).

SECONDARY OUTCOMES:
Number of patients scoring improvement of feelings using the VAS (visual analogue scale) | Baseline to 45 minutes
  We will record the number of patients scoring improvement of feelings using the VAS (visual analogue scale).

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials